CLINICAL TRIAL: NCT06224738
Title: Human HER2-targeted Chimeric Antigen Receptor Macrophages Therapy for HER2-positive Advanced Gastric Cancer With Peritoneal Metastases: an Exploratory Clinical Trial
Brief Title: Human HER2-targeted Macrophages Therapy for HER2-positive Advanced Gastric Cancer With Peritoneal Metastases
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Macera therapeutics (Unknown)
Responsible Party: Principal Investigator, Bing Xia, chief physician, First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITT-20231107-0257-02
Record Dates: First submitted 2023-12-24; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human HER2-targeted CAR-M cell (Experimental): Recombinant human granulocyte stimulating factor treatment mobilized bone marrow stem cells, when the mononuclear cells rose to more than 8×10^8/L, the collection of peripheral blood single nuclei cells, the total number of mononuclear cells collected 1.5×10^9-1.8×10^9. Intraperitoneal infusion of anti-human HER2 CAR-M cells 3×10^8 cells/person, in a single administration.According to the principle of "3+3 dose increment", enter dose 2 and dose 3. Dose2: the monocyte rises to more than 9.5×10^8/L and collect peripheral blood single nucleus cells. Reinfuse anti-human HER2 CAR-M cells 5×10^8 cells/person, 1 person/bag/dose, 100 ml/bag. Dose3: the mononuclear cell rises to more than 1.3×10^9/L and collect peripheral blood single nucleus cells. Reinfuse anti-human HER2 CAR-M cells 1×10^9 cells/person, 1 person/bag/dose, 200 ml/bag.
  Interventions: Biological: human HER2-targeted CAR-M cells

INTERVENTIONS:
Biological: human HER2-targeted CAR-M cells — The human anti-HER2 chimeric antigen receptor macrophages (anti-HER2 CAR-M cells) independently developed use adenoviral vector system to genetically engineer autologous macrophages to express CAR molecules containing single-chain antibodies, which specifically bind to the human HER2 antigen to recognize and kill tumor cells.
  Other Names: anti-HER2 CAR-M cells

SUMMARY:
The goal of this exploratory clinical trial is to evaluate the safety and efficacy of human anti-human epidermal growth factor receptor 2(HER2) Chimeric antigen receptor macrophage cells (CAR-M) in advanced HER2+ gastric cancer. Participants will mobilize bone marrow stem cells and engineer autologous macrophages to express Chimeric antigen receptor (CAR), and CAR-M will be infused intraperitoneally back into the patient for systemic anti-tumor effects.

DETAILED DESCRIPTION:
The standard approach for managing advanced peritoneal metastatic gastric cancer typically involves systemic administration of antitumor drugs. In the case of HER2-positive gastric cancer patients, a combination of trastuzumab, platinum, and fluorouracil chemotherapeutic agents is commonly employed. Nevertheless, conventional therapy encounters obstacles stemming from tumor heterogeneity and the intricate microenvironment. The self-developed humanized anti-HER2 chimeric antigen receptor macrophage (human anti-HER2 CAR-M) uses an adenoviral vector system to genetically engineer autologous macrophages to express CAR molecules containing single-chain antibodies, which specifically bind to human HER2 antigens to recognize and kill tumor cells. Cell and animal experiments as well as preclinical trials showed that anti-human HER2 CAR M cells have significant anti-tumor efficacy and good safety. This study can provide abundant clinical data for the safety and feasibility of CAR macrophage therapy for solid tumors, and promote the progress of CAR macrophage therapy for solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years (including borderline values), male or female.
2. expected survival of more than 12 weeks.
3. histologically confirmed HER2-positive gastric cancer; HER2-positive is defined as immunohistochemistry (IHC) 3+ or (IHC) 2+ with in situ hybridization (ISH) +.
4. confirmation of peritoneal metastasis by imaging or cytologic testing of peritoneal fluid.
5. presence of measurable lesions.
6. patients with peritoneal metastases of gastric cancer who had previously failed second-line or higher therapy. Treatment failure is defined as an intolerable toxic reaction or disease progression during treatment or tumor recurrence or metastasis after completion of treatment. Prior therapy of targeted agents, immunosuppressants, or radiotherapy is permitted; prior systemic therapy with at least 1-2 chemotherapeutic agents of fluorouracil, platinum, and paclitaxel in combination with targeted agents.
7. have an Eastern Cooperative Oncology Group (ECOG) activity status score of 0-2
8. at least 2 weeks have elapsed since receiving the most recent drug therapy to the time of single nucleated cell collection.
9. patients of childbearing age are required to use appropriate contraception (protection or other birth control) prior to enrollment and during the study.
10. the patient is willing to accept intraperitoneal administration of the drug.
11. the patient understands the trial and has signed an informed consent form.
12. the patient is able to follow the study protocol and follow-up procedures.

Exclusion Criteria:

1. previous or current other types of malignant tumors, except for the following: completely resected or eradicated basal and squamous cell carcinoma of the skin, and carcinoma in situ of the cervix.
2. patients requiring immunosuppressive drugs (except physiologic replacement doses).
3. history of central nervous system (CNS) disorders such as seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychosis; untreated or symptomatic CNS metastases or cytologically confirmed carcinomatous meningitis (asymptomatic CNS metastases that do not require treatment may be enrolled).
4. left ventricular ejection fraction <50%.
5. White blood cell count <3×10^9/L and platelet count <80×10^9/L.
6. AST and ALT > 3 × upper limit of normal (ULN)
7. Total bilirubin > 1.5 × ULN.
8. creatinine clearance <60 ml/min.
9. Abnormal coagulation function (activated partial thromboplastin time (APTT) > 1.5 × ULN, international normalized ratio (INR) > 1.5 × ULN).
10. patients with intestinal obstruction (gastrointestinal obstruction within 30 days prior to administration).
11. patients with infectious diseases including, but not limited to: 1) known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related disease; 2) known active liver disease, including hepatitis B and hepatitis C; 3) active tuberculosis infection, who are on anti-tuberculosis treatment or who have received anti-tuberculosis treatment within 1 year prior to the first dose of the study drug; 4) known syphilis infections requiring treatment; and 5) Other infectious diseases that, in the judgment of the investigator, make participation in this study unsuitable.
12. Diseases that, in the judgment of the investigator, preclude enrollment: including, but not limited to, severe hepatic, renal, or metabolic disease requiring drug therapy, uncontrolled coronary artery disease or asthma, and uncontrolled cerebrovascular disease.
13. pregnant or breastfeeding females; females or males of childbearing age with a pregnancy plan during the study.
14. psychotropic substance abuse, clinical or psychological or social factors that would compromise informed consent or study conduct (at the discretion of the investigator).
15. individuals who may be allergic to the study medication.
16. is participating in another clinical trial.
17. patients with inaccessible peripheral or deep venous access.
18. any uncertainty that has an impact on patient safety or compliance.
19. any other condition that the investigator considers inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse effects | The evaluation was conducted within 28 days of administration, with a total of 30 recording points
  Collect information on the type, frequency, and severity of adverse events.Identify and grade adverse events following CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Time to Sustained Remission (DOR) | 1 month, 2 months, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months post-infusion.
  Solid tumor efficacy was assessed following the RECIST 1.1 criteria, calculating the time from first onset of efficacy (i.e., complete remission (CR) or partial remission (PR)), to earliest disease progression or death.
Overall response rate (ORR) | Initiation of the first evaluation of the tumor as CR or PR to the beginning of the -th evaluation as progressive disease (PD) or death from any cause.
  Solid tumor efficacy was assessed following RECIST 1.1 criteria, and the proportion of subjects in complete or partial remission was calculated.
Disease Control Rate (DCR) | Assessed every month, up to 3 months.
  The RECIST 1.1 criteria were followed to assess the efficacy of solid tumors, and DCR was defined as the number of cases that achieved remission (CR+PR) and stable disease (SD) after treatment as a percentage of the number of evaluable cases.
Progression-free survival (PFS) | From date of administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Solid tumor efficacy was assessed following the RECIST 1.1 criteria by calculating the time between infusion and the first record of disease progression or death.
Overall Survival (OS) | From date of randomization until the date of death from any cause, assessed up to 100 months
  Calculation of time from infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xia, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Affiliated Hangzhou Cancer Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Liu L, Su H, Liu Q, Shen J, Dai H, Zheng W, Lu Y, Zhang W, Bei Y, Shen P. Chimeric antigen receptor macrophage therapy for breast tumours mediated by targeting the tumour extracellular matrix. Br J Cancer. 2019 Nov;121(10):837-845. doi: 10.1038/s41416-019-0578-3. Epub 2019 Oct 1. PMID 31570753
- [Background] Dong X, Fan J, Xie W, Wu X, Wei J, He Z, Wang W, Wang X, Shen P, Bei Y. Efficacy evaluation of chimeric antigen receptor-modified human peritoneal macrophages in the treatment of gastric cancer. Br J Cancer. 2023 Aug;129(3):551-562. doi: 10.1038/s41416-023-02319-6. Epub 2023 Jun 29. PMID 37386139